CLINICAL TRIAL: NCT03031405
Title: The Effect of Oxytocin on the Acquisition and Consolidation of Trauma-Associated Memories: A Model to Understand the Development of Posttraumatic Stress Disorder
Brief Title: The Effect of Oxytocin on the Acquisition and Consolidation of Trauma-Associated Memories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Principal Investigator, Katharina Schultebraucks, PhD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: Charite2017-Oxytocin-Study
Record Dates: First submitted 2017-01-18; First posted 2017-01-25 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2017-01

CONDITIONS: Intrusive Memories

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Oxytocin and trauma film paradigm (Experimental)
  Interventions: Drug: Oxytocin nasal spray
- Placebo and trauma film paradigm (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Oxytocin nasal spray
  Arms: Oxytocin and trauma film paradigm
Drug: Placebos — Placebo nasal spray
  Arms: Placebo and trauma film paradigm

SUMMARY:
The purpose of the study is to examine whether oxytocin and oxytocin receptor gene polymorphism affect the development of intrusive memories, a cardinal symptom of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* healthy female volunteers
* German on a native level

Exclusion Criteria:

* former or present disorder according to the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5)
* any physical illnesses
* any medication intake (except oral contraceptive)
* history of traumatic experience, e.g. history of sexual abuse or rape
* pregnancy or lactation period
* follicular phase of menstrual cycle for all women not using oral contraceptives

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Intrusive memories | four consecutive days
  Influence of oxytocin on the development of intrusive memories measured with an intrusion diary

SECONDARY OUTCOMES:
Noradrenergic System (measured with salivary alpha-amylase - u/ml) | Day 1
  Influence of oxytocin on the noradrenergic system measured with salivary alpha-amylase
Genetic polymorphism | four consecutive days
  Influence of genetic polymorphism of the oxytocin receptor on intrusive memories measured with an intrusion diary
Hypothalamic-pituitary-adrenal (HPA) axis (measured with salivary cortisol - nmol/L) | Day 1
  Influence of oxytocin on the HPA-axis measured with salivary cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Roepke, PD Dr., Study Director — Charité - Universitätsmedizin Berlin, Department of Psychiatry and Psychotherapy, Campus Benjamin Franklin
Locations (1):
- Charité - Universitätsmedizin Berlin, Department of Psychiatry and Psychotherapy, Campus Benjamin Franklin, Berlin, Germany

REFERENCES:
- [Derived] Schultebraucks K, Maslahati T, Wingenfeld K, Hellmann-Regen J, Kraft J, Kownatzki M, Behnia B, Ripke S, Otte C, Roepke S. Intranasal oxytocin administration impacts the acquisition and consolidation of trauma-associated memories: a double-blind randomized placebo-controlled experimental study in healthy women. Neuropsychopharmacology. 2022 Apr;47(5):1046-1054. doi: 10.1038/s41386-021-01247-4. Epub 2021 Dec 9. PMID 34887528